CLINICAL TRIAL: NCT03417635
Title: Meditation Strategies, Attention, and Mobility in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Lindsay Nagamatsu, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110598
Record Dates: First submitted 2018-01-12; First posted 2018-01-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Mobility Limitation
Keywords: Meditation; Cognitive assessment; Executive function; Older adults; Randomized control trial; Mobility
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided focused attention (Experimental): Participants will take part in a guided focused attention practice led by the researcher. This will include strategies used in meditations where participants focus on their breathing. More specifically, they will be instructed to close their eyes and focus on the sensation of breathing in one area of the body for the entire session. They will be given reminders throughout the session to remain on task (focusing on the breath) and not to let their thoughts wander.
  Participants will be asked to either sit on a chair or cushion on floor to ensure they are comfortable to sit still for the session, but not so much that they might fall asleep.
  Interventions: Behavioral: Guided focused attention
- Acoustic music (Active Comparator): Participants will be instructed to listen to a prepared soothing acoustic music track. The sessions will be led by a researcher. Participants will be asked to close their eyes and relax while listening to the music.
  Participants will be asked to sit on a chair or cushion on floor to ensure they are comfortable to sit still for the session, but not so much they might fall asleep This group is used as active control group to control for socialization in group settings and any effects of consciously relaxing for the meetings.
  Interventions: Behavioral: Acoustic music

INTERVENTIONS:
Behavioral: Guided focused attention — Participants will meet for 20 minute group sessions with 6-10 participants in each group. There will be three meetings a week for a four week period. The focused attention practice itself will last for 20 minutes with instructions being given during the 20 minute period. All sessions will occur in the retirement home in a community room to ensure the sessions are easily accessible to the participants.
  Arms: Guided focused attention
Behavioral: Acoustic music — Participants will meet for 20 minute group sessions with 6-10 participants in each group. There will be three meetings a week for a four week period. The acoustic music track itself will last for 20 minutes with instructions being given during the 20 minute period. All sessions will occur in the retirement home in a community room to ensure the sessions are easily accessible to the participants.
  Arms: Acoustic music

SUMMARY:
Approximately 30% of community-dwelling older adults experience one or more falls per year, resulting in injuries, loss of independence, and reduced quality of life. While there are known physiological risk factors for falls, including poor balance and altered gait patterns, it is now recognized that impaired cognitive functioning is also a risk factor for falls. Within the broad construct of cognition, one specific domain that has been focused on in the falls literature is attention. The literature suggests that improving attention in those at-risk for falls may reduce older adult's risk of falling.

DETAILED DESCRIPTION:
The current study aims to investigate the impact of meditation strategies on measures of attention and electrical signals in the brain in older adults. Investigators will recruit older adults who are living in the community. Participants will be assigned to one of two groups: 1) guided focused attention group, or 2) music group (control group). All participants will complete three in-person sessions per week and then be encouraged to practice independently on the other days in the week, for a total of four weeks.The current study focuses on focused attention meditation strategies, as it is recommended for beginner-level meditators. This will include training to be able to focus on one's breathing for 20 minute sessions. Focused attention meditation has been found to increase levels of executive functioning and attention. Participants will complete mobility and cognitive assessments at both the beginning and end of the intervention. These will be completed in the retirement homes for convenience. Participants will also attend an in-lab session to complete electroencephalogram (EEG) testing at both timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. minimum 60 years of age,
2. minimum completed high school,
3. must be comfortable writing and reading English,
4. be able to walk independently,
5. must be right-handed (for EEG analysis),
6. score 6+/8 on the instrumental activities of daily living scale,
7. score >24/30 on the Mini-Mental Status examination.

Exclusion Criteria:

To be included, participants must NOT:

1. have a diagnosis of neurodegenerative disease,
2. have a diagnosis of cognitive impairment (e.g., MCI),
3. have a diagnosis of a psychiatric condition,
4. have had a concussion in the last 12 months,
5. have had a stroke,
6. have musculoskeletal or joint disease,
7. experience dizziness or loss of balance,
8. have visual, auditory, or somatosensory impairment, or
9. a recent history (past 2 years) of regular meditation practice (1 or more times per week) or include a meditation component in their religious practice.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in sustained attention | 4 weeks
  Measured by performance on sustained attention task.

SECONDARY OUTCOMES:
Change in global attention | 4 weeks
  Measured by electrophysiological measures of attention.
Change in mobility | 4 weeks
  Measured by the Timed Up and Go test.
Change in mobility and balance | 4 weeks
  Measured by the Short Physical Performance Battery.
Change in memory | 4 weeks
  Measured with the Rey Auditory Verbal Learning Test
Change in conflict resolution | 4 weeks
  Measured with the stroop task
Change in set-shifting | 4 weeks
  Measured with the trail making task
Change in working memory | 4 weeks
  Measured with the digit span task

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay S Nagamatsu, PhD, Principal Investigator — Western University
Locations (1):
- Community, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin K, Thomson R, Blizzard L, Wood A, Garry M, Srikanth V. Visuospatial ability and memory are associated with falls risk in older people: a population-based study. Dement Geriatr Cogn Disord. 2009;27(5):451-7. doi: 10.1159/000216840. Epub 2009 May 7. PMID 19420939
- [Background] Nagamatsu LS, Liu-Ambrose TY, Carolan P, Handy TC. Are impairments in visual-spatial attention a critical factor for increased falls risk in seniors? An event-related potential study. Neuropsychologia. 2009 Nov;47(13):2749-55. doi: 10.1016/j.neuropsychologia.2009.05.022. Epub 2009 Jun 6. PMID 19501605
- [Background] Nagamatsu LS, Munkacsy M, Liu-Ambrose T, Handy TC. Altered visual-spatial attention to task-irrelevant information is associated with falls risk in older adults. Neuropsychologia. 2013 Dec;51(14):3025-32. doi: 10.1016/j.neuropsychologia.2013.10.002. PMID 24436970
- [Background] Wallace, B. A. (2006). The attention revolution: Unlocking the power of the focused mind. Somerville, Massachusetts: Wisdom Publications, Inc.
- [Background] Ainsworth B, Eddershaw R, Meron D, Baldwin DS, Garner M. The effect of focused attention and open monitoring meditation on attention network function in healthy volunteers. Psychiatry Res. 2013 Dec 30;210(3):1226-31. doi: 10.1016/j.psychres.2013.09.002. Epub 2013 Oct 14. PMID 24135553
- [Background] Tsai MH, Chou WL. Attentional orienting and executive control are affected by different types of meditation practice. Conscious Cogn. 2016 Nov;46:110-126. doi: 10.1016/j.concog.2016.09.020. Epub 2016 Oct 3. PMID 27710818
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Ford SD, Nagamatsu LS. Four weeks of meditation training improves sustained attention in community-dwelling older adults: a proof-of-concept randomized controlled trial. Front Aging. 2024 Mar 1;5:1322705. doi: 10.3389/fragi.2024.1322705. eCollection 2024. PMID 38496316
- [Derived] Nagamatsu LS, Ford SD. Can meditation improve attention in older adults? Study protocol for a 4-week proof-of-concept intervention. Pilot Feasibility Stud. 2019 Feb 11;5:22. doi: 10.1186/s40814-019-0413-x. eCollection 2019. PMID 30788136